CLINICAL TRIAL: NCT00266175
Title: Pulmonary Arteriopathy; Evaluation of Invasive Treatments of Peripheral Pulmonary Stenosis in Terms of Right Ventricular Function and Patient Exercise Tolerance
Brief Title: Pulmonary Arteriopathy-Diagnostics and Therapy
Status: Completed | Type: Observational
Sponsor: Competence Network for Congenital Heart Defects (Other Government)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Other Study IDs: MP 1; 01G10210
Record Dates: First submitted 2005-12-15; First posted 2005-12-16 (Estimated); Last update posted 2008-10-15 (Estimated); Status verified 2008-10

CONDITIONS: Pulmonary Stenosis
Keywords: Pulmonary heart disease; Pulmonary hypertension; Stent implantation; Balloon dilatation; Surgery
MeSH Terms: conditions — Pulmonary Valve Stenosis; Pulmonary Heart Disease; Hypertension, Pulmonary

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Postoperative stenoses of the pulmonary artery vascular system seldom occur alone; they are frequently found in connection with congenital heart defects or malformation syndromes. The resulting increase of afterload represents a serious pressure load for the right ventricle. Depending on the number and severity of the stenoses, gradual functional right ventricular failure is to be expected. Due to limited clinical experience, there has not yet been a consensus concerning the indications for the different therapeutic strategies (balloon dilatation, stent implantation, surgical dilatation techniques). Up to now, only few investigators in few centres use stents as therapy. Therefore, systematic multicenter investigations assessing larger groups of patients undergoing this procedure are not yet available. The same applies to other novel dilatation techniques, such as the use of the "cutting balloon" as therapy for rigid valve stenoses.

By comparing and analysing different invasive forms of treatment (balloon dilatation, stent implantation and surgery), we expect to achieve an optimisation of therapy.

In the study, the outcomes of different strategies as practiced now in German cardiological centers will be compared and the main factors influencing the results will be determined. On the basis of a standardized investigation before and one year after the intervention, these comparisons with respect to the reduction of stenosis and corresponding changes of right ventricular functional and anatomical changes are carried out correcting for known confounders. The assessment of the different included invasive and non-invasive diagnostical procedures with respect to their ability to detect pathological findings and their changes as result of the treatment is an important secondary target of the study.

DETAILED DESCRIPTION:
For patients with untreated peripheral pulmonary stenoses, the course of disease is characterised by a chronic pressure load of the right ventricle. In the medium to long term this can lead to right heart failure and cardiac arrhythmia unresponsive to therapy. The probability of these events as well as the time of their occurrence depends on the severity of the stenoses, the duration of stress and a possible additional volume load. Within the scope of the prospective study introduced here, we intend to characterise the stenoses with respect to degree and type and to document the treatment success in terms of decrease of afterload of the right ventricle. In this context, imaging and catheter-based methods as well as respective functional analyses are to be used to provide evidence of a reduction or neutralisation of the pulmonary artery stenoses.

Accordingly, the following questions, or corresponding objectives, can be identified as the base for the conduct of this clinical trial:

* Morphological and functional categorisation of the angiostenoses and standardisation of the diagnostic procedures. For this purpose, the quantitative criteria for both the morphological degree of stenosis (lumen constriction) and the functional degree of stenosis (pressure gradient) are established by means of cardiac catheterisation and angiography. Non-invasive imaging methods, which have as yet been restricted primarily to echocardiography, are complemented by the method of spin angiography. Compared to conventional angiography, this has the advantage of being less invasive and not involving radiation exposure.
* On the strength of past experience, the implantation of stents can be viewed as a very promising approach to a treatment with lasting effectiveness of pulmonary artery stenoses. The stents have the advantage of high radial forces that can be offset against the elastic recoil of the vessels occurring after sole dilatation. Furthermore, constrictions that are caused by either kinking of vessels or their compression by neighbouring structures can be dilated sufficiently by the use of stents.
* With respect to the interconnectedness of all the projects of the Competence Network for Congenital Heart Defects, one essential aspect is the standardisation of diagnostic methods of evaluating right ventricular function. The data obtained during the study are to provide the basis for the development of diagnostic guidelines.
* Concerning evaluation, particular attention is paid to the patients' self-assessment with respect to their exercise tolerance. In this context, it is a matter of interest to what degree the patients' subjective maximum stress and therefore their quality of life correlate with the objective measurement parameters. The anticipated results are of direct clinical significance for the patients, as they aim at medium to long-term relief of the right ventricle, which may effect a decrease in morbidity and therefore an improvement of the quality of life. This is of particular importance with regard to the fact that there will be a continuously increasing number of patients with congenital heart defects reaching adulthood.

ELIGIBILITY:
Inclusion Criteria:

Patients with native or postoperative peripheral pulmonary stenoses (PPS; any stenoses that are located distally to the RVOT). Definition of PPS: 40% lumen constriction, or 30% constriction if volume stress is also present. Informed consent of the patient or his/her legal representative is given after instruction. -

Exclusion Criteria:

Patients unable to undergo MRI or spiroergometry for physical or psychological reasons.

Pregnant or nursing patients. Patients affected by other clinically relevant diseases (malignant tumours, infectious diseases, metabolic disorders etc.). Patients with known intolerance of contrast media. Patients with syndromal diseases such as Alagille's syndrome, rubella embryopathy or elfin face syndrome. -

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2005-05; Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Primary outcome measure:
To assess the efficacy of the administered therapy, both the ectasia of the stenosed vessels in
relation to the target diameter and the reduction of the pressure gradient in the stenosed vessel
are indicated in percent. An evaluation of the therapeutic success takes place after twelve months.
Definition of the primary target of therapy:
Morphometric:
• Expansion of the peripheral pulmonary artery stenosis to at least 80% of the vascular
lumen.
Manometric:
• Gradient reduction over the stenosis of at least 50%.
• Reduction in right ventricular systolic pressure, indicated by a reduced ratio of systolic
pressure of LV to RV. In this context, there is no definition in terms of a primary target,
as right ventricular pressure reduction depends on a variety of parameters (such as
number of stenoses of the entire peripheral pulmonary vasculature, potential
additional volume load and right ventricular overall function).

SECONDARY OUTCOMES:
Secondary outcome measures:
The improvement of the right ventricular systolic and diastolic function as well as reduction of
ventricle size and of tricuspid valve incompetence are quantified by means of echocardiography,
angiography and, where required, nuclear magnetic resonance tomography.
An improvement in capability/quality of life is assessed by means of bicycle ergometer
examinations as well as the SF-36 (New England Hospital Inc.) and KINDL questionnaires
(Ravens-Sieberer & Bullinger) for adults and children respectively.
In assessing the organ-related outcome measures, the different diagnostic imaging methods are
compared with each other.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Schneider, MD, Principal Investigator — Deutsches Kinderherzzentrum
Locations (5):
- Germany (5):
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Herz-und Diabeteszentrum NRW, Bad Oeynhausen, North Rhine-Westphalia
  - Deutsches Kinderherzzentrum, Sankt Augustin, North Rhine-Westphalia
  - Universitätsklinikum des Saarlandes, Homburg, Saarland
  - Deutsches Herzzentrum Berlin, Berlin, State of Berlin